# **Signature Page**

# Safety Evaluation of an Advanced Hybrid Closed Loop System Using Lyumjev with the Tandem t:slim X2 with Control-IQ in Adults, Adolescents and Children with Type 1 Diabetes

Protocol Identifying Number: TP-0009650 IDE Sponsor: Tandem Diabetes Care, Inc.

Version Number: v. 4.0 13 APR 2022

| Sponsor | |
|-----------------|----------------------|
| Name, degree | Jordan Pinsker, MD |
| Signature/Date | |
| Sponsor | |
| Name, degree | John W. Lum, MS |
| Signature/Date | |
| Medical Monitor | |
| Name, degree | Roy W. Beck, MD, PhD |
| Signature/Date | |

Safety Evaluation of an Advanced Hybrid Closed Loop System Using Lyumjev with the Tandem t:slim X2 with Control-IQ in Adults, Adolescents and Children with Type 1 Diabetes

Protocol Identifying Number: TP-0009650 IDE Sponsor: Tandem Diabetes Care, Inc.

Version Number: v. 4.0 13 APR 2022

# **KEY ROLES**

| Sponsor and Clinical Director | |
|-----------------------------------|-------------------------------------|
| Name, degree | Jordan Pinsker, MD |
| Title | Vice President and Medical Director |
| Institution Name | Tandem Diabetes Care, Inc. |
| JCHR Coordinating Center Director | |
| Name, degree | John W. Lum, MS |
| Title | Coordinating Center Director |
| Institution Name | Jaeb Center for Health Research |
| Medical Monitor | |
| Name, degree | Roy W. Beck, MD, PhD |
| Title | Medical Director |
| Institution Name | Jaeb Center for Health Research |

# TABLE OF CONTENTS

| CHAPTER 1: BACKGROUND INFORMATION | 16 |
|---------------------------------------------------------|----|
| 1.1 Introduction | 16 |
| 1.1.1 Tandem X2 Insulin Pump with Control-IQ Technology | 16 |
| 1.1.2 Lyumjev Insulin | 16 |
| 1.2 Rationale | 17 |
| 1.3 Potential Risks and Benefits | 17 |
| 1.3.1 Known Potential Risks | 17 |
| 1.3.1.1 Blood Draw | 17 |
| 1.3.1.2 CGM and Pump Catheter Risks | 17 |
| 1.3.1.3 Hypoglycemia | 17 |
| 1.3.1.4 Risk of Hyperglycemia | 18 |
| 1.3.1.5 Risk of Device Reuse | 18 |
| 1.3.1.6 Questionnaires | 18 |
| 1.3.1.7 Potential Risks of the CLC System | 18 |
| 1.3.1.8 Potential Risks of Using Lyumjev | 18 |
| 1.3.1.9 Other Risks. | 19 |
| 1.3.2 Benefits | 19 |
| 1.3.3 Risk Assessment | 19 |
| 1.4 General Considerations. | 19 |
| CHAPTER 2: STUDY ENROLLMENT AND LEAD-IN PERIOD | 20 |
| 2.1 Participant Recruitment and Enrollment | 20 |
| 2.1.1 Informed Consent and Authorization Procedures | 20 |
| 2.2 Participant Eligibility Criteria | 21 |
| 2.2.1 Inclusion Criteria | 21 |
| 2.2.2 Exclusion Criteria | 22 |
| 2.3 Screening Procedures | 23 |
| 2.3.1 Data Collection and Testing | 23 |
| 2.4 Screen Failures | 23 |
| 2.5 Lead-in Period | 24 |
| CHAPTER 3: TREATMENT PERIOD | 25 |
| 3.1 CIQ 1.5/ Lyumjev Training Visit | 25 |
| 3.1.1 Training on System Use | 25 |
| 3.1.2 Training on Management of Hypoglycemia | 26 |
| 3.1.3 Training on Management of Hyperglycemia | 26 |

| 3.1.4 Participant Reporting of Infusion Set Insertion Reactions | 27 |
|---|---|
| 3.1.5 Adjustments in Insulin Pump Settings | 27 |
| 3.2 Study Visits and Phone Contacts | 27 |
| 3.2.1 Procedures During Phone Contacts | 27 |
| 3.2.2 Procedures at Study Visits | 28 |
| 3.2.3 Unscheduled Visits | 28 |
| 3.3 Exercise and Meal Challenges | 28 |
| Participants will complete 3 meal and 3 exercise challenges during Lyumjev use. Procedures are described in section 5.1. | 28 |
| 3.4 Early Discontinuation of Study Device | 28 |
| CHAPTER 4: STUDY DEVICES AND DRUGS | 29 |
| 4.1 Study Devices | 29 |
| 4.1.1 Insulin Pump. | 29 |
| 4.1.2 Continuous Glucose Monitoring | 29 |
| 4.1.3 Blood Glucose Meter | 29 |
| 4.1.4 Ketone Meter | 29 |
| 4.2 Study Drug. | 29 |
| 4.3 Study Device and Drug Accountability Procedures | 30 |
| 4.4 Participant Access to Study Device at Study Closure | 30 |
| CHAPTER 5: TESTING PROCEDURES AND QUESTIONNAIRES | |
| 5.1 Meal and Exercise Challenges | |
| 5.1.1 Meal Challenges | |
| 5.1.2 Exercise Challenges. | |
| 5.2 Laboratory Testing | |
| 5.2.1 HbA1c | |
| 5.2.2 Urine Pregnancy | |
| 5.3 Questionnaires | 33 |
| CHAPTER 6: UNANTICIPATED PROBLEM, ADVERSE EVENT, AND DEVICE ISSUE REPORTING | |
| 6.1 Unanticipated Problems | |
| 6.2 Adverse Events | |
| 6.2.1 Definitions | |
| 6.2.2 Reportable Adverse Events | |
| 6.2.3 Hypoglycemic Events | |
| 6.2.4 Hyperglycemic/Ketotic Events | |
| 6.2.5 Skin Reactions Related to Infusion Set | |
| 6.2.6 Relationship of Adverse Event to Study Investigational Device | 37 |

| 6.2.7 Severity (Intensity) of Adverse Events | 37 |
|-----------------------------------------------------------------|----|
| 6.2.8 Expectedness | 38 |
| 6.2.9 Coding of Adverse Events | 38 |
| 6.2.10 Outcome of Adverse Events | 38 |
| 6.3 Reportable Device Issues | 39 |
| 6.4 Timing of Event Reporting | 39 |
| 6.5 Safety Oversight | 40 |
| 6.6 Stopping Criteria | 40 |
| 6.6.1 Participant Discontinuation of Study Device | 40 |
| 6.6.2 Criteria for Suspending or Stopping Overall Study | 41 |
| CHAPTER 7: MISCELLANEOUS CONSIDERATIONS | |
| 7.1 Drugs Used as Part of the Protocol | |
| 7.2 Collection of Medical Conditions and Medications | 42 |
| 7.3 Prohibited Medications, Devices, Treatments, and Procedures | 42 |
| 7.4 Rescue Medications, Treatments, and Procedures | 42 |
| 7.5 Pregnancy Reporting | 42 |
| 7.6 Participant Compensation | 42 |
| 7.7 Participant Withdrawal | 42 |
| 7.8 Confidentiality | 43 |
| CHAPTER 8: STATISTICAL CONSIDERATIONS | 44 |
| 8.1 Statistical and Analytical Plans | 44 |
| 8.2 Statistical Hypotheses | 44 |
| 8.3 Sample Size | 44 |
| 8.4 Outcome Measures | 44 |
| 8.5 Analysis Datasets | 45 |
| 8.6 Statistical Methods | 45 |
| 8.6.1 Analysis of the Safety Event Endpoints | 45 |
| 8.6.2 Analysis of CGM Endpoints | 45 |
| 8.6.3 Analysis of HbA1c and PRO Measures | 45 |
| 8.7 Intervention Adherence | 46 |
| 8.8 Protocol Adherence and Retention | 46 |
| 8.9 Baseline Descriptive Statistics | 46 |
| 8.10 Additional Tabulations and Analyses | 46 |
| 8.11 Device Issues | 47 |
| 8.12 Planned Interim Analyses | 47 |
| 8.13 Subgroup Analyses | 47 |

| 8.14 Multiple Comparison/Multiplicity | 47 |
|-----------------------------------------------------|----|
| 8.15 Analysis of Meal and Exercise Challenges | 47 |
| CHAPTER 9: DATA COLLECTION AND MONITORING | 48 |
| 9.1 Case Report Forms and Other Data Collection | 48 |
| 9.2 Study Records Retention | 48 |
| 9.3 Quality Assurance and Monitoring | 48 |
| 9.4 Protocol Deviations | 49 |
| CHAPTER 10: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 50 |
| 10.1 Ethical Standard | 50 |
| 10.2 Institutional Review Boards | 50 |
| 10.3 Informed Consent Process | 50 |
| 10.3.1 Consent Procedures and Documentation | 50 |
| 10.3.2 Participant and Data Confidentiality | 50 |
| 10.3.3 Future Use of Stored Specimens and Data | 51 |
| Chapter 11: References | 52 |

# **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|--------------|-----------------------------------------------|
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| BGM | Blood Glucose Meter |
| BMI | Body Mass Index |
| CFR | Code of Federal Regulations |
| CGM | Continuous Glucose Monitoring |
| DCCT | Diabetes Control & Complications Trial |
| DKA | Diabetic Ketoacidosis |
| eCRF | Electronic Case Report Form |
| GCP | Good Clinical Practice |
| HbA1c | Hemoglobin A1c |
| ICH | International Conference of Harmonization |
| IDE | Investigational Device Exemption |
| IRB | Institutional Review Board |
| RBM | Risk-Based Monitoring |
| SAE | Serious Adverse Event |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| T1D | Type 1 Diabetes |
| UADE | Unanticipated Adverse Device Effect |

### SITE PRINCIPAL INVESTIGATOR STATEMENT OF COMPLIANCE

Protocol Title: Safety Evaluation of an Advanced Hybrid Closed Loop System Using Lyumjev with the Tandem t:slim X2 with Control-IQ in Adults, Adolescents and Children with Type 1 Diabetes

Protocol Version/Date: 4.0 13 APR 2022

I have read the protocol specified above. In my formal capacity as a Site Principal Investigator, my duties include ensuring the safety of the study participants enrolled under my supervision and providing the Jaeb Center for Health Research, which serves as the Coordinating Center for the protocol, with complete and timely information, as outlined in the protocol. It is understood that all information pertaining to the study will be held strictly confidential and that this confidentiality requirement applies to all study staff at this site.

This trial will be carried out in accordance with ICH E6 Good Clinical Practice (GCP) and as required by the following: United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812).

Also, the trial will be carried out in accordance with ICH E6 Good Clinical Practice (GCP), and the Declaration of Helsinki.

As the Principal Investigator, I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), or other approved Ethics Committee, except where necessary to eliminate an immediate hazard(s) to the trial participants.

All key personnel (all individuals responsible for the design and conduct of this trial) have completed Human Participants Protection Training and Good Clinical Practice Training. Further, I agree to ensure that all staff members involved in the conduct of this study are informed about their obligations in meeting the above commitments.

| Investigator's Signature | Date: | | / / | |
|--------------------------|-------|----|-----|------|
| | | dd | mmm | уууу |
| Investigator's Name: | | | | |
| Site Name/Number: | | | | |

# PROTOCOL SUMMARY

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Study Sponsor | Tandem Diabetes Care, Inc. |
| Protocol Number | TP-0009650 |
| Protocol Title | Safety Evaluation of an Advanced Hybrid Closed Loop System Using Lyumjev with the Tandem t:slim X2 with Control-IQ in Adults, Adolescents and Children with Type 1 Diabetes |
| Précis | This is a prospective, multi-center (US only), single-arm study in adults and children (ages 6 to <81 years) with type 1 diabetes (T1D) who are current users of the t:slim X2 pump with Control-IQ technology to evaluate the safety of Lyumjev in the Control-IQ 1.5 System to achieve labeling updates for Lyumjev and the t:slim X2 insulin pump with Control-IQ 1.5 technology. Participants will be current Control-IQ users who will use Humalog with the study pump (Control-IQ 1.5) during a ~16 day lead-in during which pump setting adjustments may be made in response to observed trends. This will be followed by a 3-month outpatient treatment period in which participants will use the study pump with Control-IQ 1.5 and Lyumjev insulin. |
| | Exercise and meal challenges will be performed during the lead-in period and the main study period. |
| Products | Hybrid Closed Loop System: |
| | • t:slim X2 pump with Control-IQ 1.5 technology |
| | Dexcom G6 system |
| | Lyumjev (insulin lispro-aabc) |
| Objectives | To evaluate the safety of Lyumjev (insulin lispro-aabc) use in the Tandem t:slim X2 insulin pump with Control-IQ 1.5 technology in adult and pediatric participants with diabetes in an outpatient setting to support system labeling. |
| Number of Sites | ~10-15 clinical sites in the US. |
| Study Design | Single-arm prospective safety trial |
| Number of Participants | Up to 200 participants commencing treatment period so that at least 160 complete study (at least 80 participants age 6-<14 years old, and at least 80 participants age 14+). At least 20 participants will be age 14-<18 years of age. |
| | <ul> <li>Goal to have at least 1/3 of all completers with HbA1c ≥7.5%</li> </ul> |
| | • Goal to have at least 10 completers with basal insulin rate >3 units/hour (for at least part of the day) |
| | Enrollment will be staged, starting with the 14+ cohort. After a cumulative 10,000 hours of use are reached in the age 14+ cohort, a Trial Level Safety Review of all adverse events and device issues will be performed before opening enrollment to the 6-13 year old cohort. |
| Participant Population: | Eligibility to enroll in the study will be assessed based on the following inclusion criteria: |
| | 1. Age 6 to <81 years |
| | 2. Diagnosis of type 1 diabetes for at least 1 year |
| | 3. Currently using Control-IQ technology for at least 3 months, with system use (active closed loop) for at least 85% of the possible time in 14 days prior to enrollment |
| | 4. Total daily insulin dose (TDD) at least 2 U/day |
| | 5. $HbA1c < 10.5\%$ |
| | 6. Residing full-time in the United States, with no anticipated travel outside the United States during the period of study participation. |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | <ul> <li>7. For participants &lt;18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia, able to contact the participant in case of an emergency, and willing to use the Dexcom Follow app (with push notifications turned on) for the duration of the study.</li> <li>8. If &gt;18 years old, participant has someone who lives within 30 minutes of them who is willing to be contacted if the study team can't reach the participant in case</li> </ul> |
| | <ul> <li>of a suspected medical emergency.</li> <li>9. Participant has agreed to participate in the study; and has read, understood and signed the informed consent form (ICF) and assent, if applicable; and has agreed to follow all study procedures, including:</li> </ul> |
| | <ul> <li>suspending use of any personal CGM for the duration of the clinical trial once the study CGM is in use</li> <li>switching to or continuing to use Humalog during the lead-in period</li> <li>switching to Lyumjev for the main study period.</li> </ul> |
| | willing and able to perform the study exercise and meal challenges. |
| | 10. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, including ability to respond to alerts and alarms, and to provide basic diabetes self-management. |
| | <ol> <li>Participant and/or parent/legal guardian have the ability to read and understand<br/>English</li> </ol> |
| | Eligibility to enroll in the study will be assessed based on the following exclusion criteria: |
| | 1. More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months |
| | 2. More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months |
| | 3. Inpatient psychiatric treatment in the past 6 months |
| | 4. History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to screening or unwillingness to agree to abstain from illicit drugs throughout the study. |
| | 5. For Female: Currently pregnant or planning to become pregnant during the time period of study participation |
| | <ul> <li>A negative pregnancy test will be required for all females of child-bearing<br/>potential (menarchal)</li> </ul> |
| | <ul> <li>Counseling on appropriate birth control options will be provided to females<br/>with child-bearing potential in the event the participant does not have an<br/>acceptable plan.</li> </ul> |
| | 6. Adults lacking the capacity to provide consent and/or follow study procedures in the opinion of the investigator |
| | 7. Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas). |
| | 8. Hemophilia or any other bleeding disorder |
| | 9. Hemoglobinopathy |
| | <ol> <li>History of heart, liver, lung or kidney disease determined by investigator to<br/>interfere with the study</li> </ol> |
| | 11. History of allergic reaction to Humalog or Lyumjev |
| | <ol> <li>Use of glucocorticoids, beta blockers or other medications determined by<br/>investigator to interfere with study</li> </ol> |
| | 13. Abnormal screening electrocardiogram consistent with increased risk during exercise, such as arrhythmia, ischemia, or prolonged QTc interval (>450 ms) |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | (Screening ECG only required for participants age > 50, duration of diabetes > 20 years, or history of coronary artery disease) |
| | <ol> <li>Significant chronic kidney disease (which could impact CGM accuracy in<br/>investigator's judgment) or hemodialysis</li> </ol> |
| | 15. History of adrenal insufficiency |
| | <ol> <li>History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that<br/>is not appropriately treated</li> </ol> |
| | 17. History of gastroparesis |
| | <ol> <li>A condition, which in the opinion of the investigator or designee, would put the<br/>participant or study at risk</li> </ol> |
| | <ol> <li>Participation in another pharmaceutical or device trial at the time of enrollment or<br/>anticipated for during the time period of study participation</li> </ol> |
| | 20. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., Eli Lilly and Co., or TypeZero Technologies, LLC, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial |
| Participant Duration | Approximately 15 weeks (~16 days for run in period followed by 13 weeks of study device use with Lyumjev). |
| Study Endpoints | The adult and pediatric populations will be combined for primary analysis. Separate secondary analyses also will be performed for the adult and pediatric cohorts. CGM metric analyses will be analyzed separately for the challenge days and subsequent nights and not included in the overall analyses. |
| | Primary Safety Endpoints: |
| | <ul> <li>Severe hypoglycemia (with cognitive impairment such that assistance of another<br/>individual is needed for treatment) during study compared with data on severe<br/>hypoglycemic events reported by T1D Exchange clinic registry over a 3-month time<br/>period.</li> </ul> |
| | Diabetic ketoacidosis |
| | Unanticipated adverse device effects |
| | Other serious adverse events |
| | Adverse drug reactions |
| | Secondary Safety Endpoints: |
| | All adverse events (including infusion site reactions) |
| | <ul> <li>CGM hypoglycemia outcomes (compared with baseline run-in data and separately<br/>when possible with 4 weeks of pre-study CGM data collected at enrollment)</li> </ul> |
| | ◆ Overall % time <54 mg/dL |
| | • Postprandial % time $<54$ mg/dL (30 min, $\le1$ , $\le2$ , $\le4$ , $>1$ to $\le2$ and $>2$ to $\le4$ hr) |
| | • Overall and postprandial % time <70 mg/dL |
| | <ul> <li>Rate of hypoglycemia events defined as 15 or more consecutive minutes</li> <li>4 mg/dL</li> </ul> |
| | Exploratory: |
| | Postprandial incremental area under the glucose curve (4 hr) |
| | Peak postprandial glucose The state of the state of |
| | • Times in ranges-overall and postprandial (70-180 mg/dL, >180 mg/dL, >250 mg/dL, 70-140 mg/dL) |
| | Mean glucose |
| | <ul> <li>Rate of hyperglycemia events, defined as 90 or more minutes &gt;300 mg/dL within<br/>120 minutes</li> </ul> |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | Overall variability (CV and SD) |
| | HbA1c change from baseline |
| | Patient-reported outcomes |
| | Exercise and Meal Challenges: |
| | <ul> <li>Endpoints will be CGM metrics and safety outcomes as indicated above</li> </ul> |
| | Separate analyses conducted for the overnight following the challenge |
| Protocol Overview/Synopsis | After consent is obtained, eligibility will be assessed. Eligible participants will enter the Lead-in Period. |
| | <u>Lead-in Period</u> : |
| | The lead-in Period will last approximately 16 days, and may begin the same day the screening visit is completed. Participants will switch from their current Control-IQ system to the study pump (Control-IQ 1.5 technology) and study sensor, and will be trained by qualified study staff on the new study devices including use of Humalog (insulin lispro injection). Study participation will require use of the Control-IQ technology with at least 85% of active closed loop over ~16 days of the lead-in period. The lead-in period data collection may be repeated if this threshold is not met. |
| | A study meal challenge and exercise challenge will be performed with Humalog during the lead in period. Those day and overnight periods will be analyzed separately. |
| | Treatment Period: |
| | Participants will return to clinic to undergo device training with Lyumjev in the study pump. |
| | Participants will then use the study pump and the investigational insulin for ~90 days during the study period. Participants will have a phone follow up visit at 1 week and 3 weeks, a clinic follow up visit at 6 weeks, a phone follow up visit at 9 weeks, and a final clinic visit at ~13 weeks. |
| | Participants will use the t:slim X2 insulin pump with Control-IQ technology turned on with the investigational insulin. It is acceptable to use manual mode when there is a loss of CGM data. |
| | Weekly phone/email/text contacts will be performed as part of the comprehensive plan to monitor for adverse events, to include infusion site reactions. |
| | Each participant will perform 3 meal and 3 exercise challenges during Lyumjev use. |
| | An assessment of adverse events, using open ended questions to capture hyperglycemic and hypoglycemic events, and their underlying cause and relationship to the study device, study insulin or other parts of the system (such as the infusion set), will occur at all visits/contacts. Study Safety Plan: |
| | Participants will be given a blood glucose and ketone meter to use throughout the study, and will be trained on their use by qualified staff. BGM readings will be performed in accordance with the study safety plan and per CGM manufacturer instructions. Ketone readings will be performed per the study safety plan. |
| | Site investigators may adjust insulin delivery profile settings as needed throughout the study in accordance with their clinical practice. |

## **SCHEMATIC OF STUDY DESIGN**



| | Screening<br>Visit | CIQ 1.5/<br>Humalog<br>Training<br>Visit | CIQ 1.5/<br>Lyumjev<br>Training<br>Visit | Control-IQ Use | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Lead-In | Start Main<br>Trial<br>~16 days<br>after start<br>of Lead-In | 3d | 1w | 2w | 3w | 6w | 9w | 13w | UV |
| Visit (V) or Contact (C) | V | V | V | C | C | C | C | V | C | V | V/C |
| Informed Consent/Assent | X | | | | | | | | | | |
| Eligibility Assessment | X | | | | | | | | | | |
| Medical history/<br>physical exam <sup>a</sup> | X | | | X | X | X | X | X | X | X | X |
| Height, weight,<br>blood pressure and pulse | X | | X | | | | | | | | |
| HbAlc (POC or local lab) | X | | | | | | | | | | |
| ECG <sup>b</sup> | X | | | | | | | | | | |
| Questionnaires/Surveys<br>(PRO Assessments) <sup>c</sup> | X | | | | | | | | | X | |
| Pregnancy test (females of child-bearing potential) | X | | X | | | | | | | | |
| Assessment of Device Use | X | | X | | | | | | | | |
| Study system training | | X | X | | | | | | | | |
| HbA1c (Central Lab) | | | X | | | | | | | X | |
| AE Assessment | | X | X | X | X | X | X | X | X | X | X |
| Upload device data from home | | | | X | X | X | X | | X | | X |
| Download device data at clinic visit | X | X | X | | | | | X | | X | X |

<sup>&</sup>lt;sup>a</sup> A qualified medical professional must perform a medical assessment at each office visit. During each office visit, the skin

9

10

<sup>5</sup> surrounding the infusion sites should be assessed as part of a focused physical exam. This also applies for all phone visits

<sup>6</sup> converted to an office visit, as well as unscheduled visits that occur in the office.

<sup>&</sup>lt;sup>b</sup> ECG performed at screening for participants age >50 years, duration of diabetes > 20 years, or history of coronary artery disease

<sup>8 °</sup> TRIM-D, Trim-DD (Diabetes Device), ITSQ (Insulin Treatment Satisfaction Questionnaire)

# **Chapter 1: Background Information**

#### 1.1 Introduction

#### 1.1.1 Tandem X2 Insulin Pump with Control-IQ Technology

The Tandem X2 insulin pump with Control-IQ technology is an FDA-approved closed-loop control (CLC) system based on the control algorithm developed and initially tested in the University of Virginia's DiAs system and then implemented in the inControl system (TypeZero, Technologies, Inc.). Use of the Control-IQ system has been extensively tested in adults and children with type 1 diabetes (T1D), demonstrating its efficacy and safety when used with insulin lispro (Humalog) or insulin aspart (Novolog). The system is currently approved for ages 6 years and older and it is use in younger children is currently being studied (clinical trials.gov NCT04796779). There are over 150,000 users of the system since it became commercially available in 2020. A recent evaluation of real-world use of the system in 9,451 users age  $\geq$ 6 years with at least 12 months of system use found results comparable to those found in the randomized trials.<sup>3</sup>

Since the initial approval of the system, modifications have been made in the software, which is referred to as version 1.5. These modifications include modest usability improvements and other enhancements intended to further reduce risk.

#### 1.1.2 Lyumjev Insulin

Lyumjev<sup>TM</sup> is a rapid-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. It has a faster onset of action and shorter duration of action than Humalog® (insulin lispro). Insulin lispro appears in the bloodstream approximately 1 minute after injection of Lyumjev, 5 minutes faster than Humalog. In pharmacodynamic euglycemic clamp studies comparing Lyumjev and Humalog, onset of action was 10-min faster and duration of action was 44 minutes shorter with Luymjev compared to Humalog across all populations and dose range.<sup>4</sup> Lyumjev may be given as part of a multiple daily insulin regimen or administered via continuous subcutaneous insulin infusion. This is the first clinical trial evaluating Lyumjev with Control-IQ technology.



- 40 The differences in insulin lispro PK profiles between LY900014 and Humalog following SC injection
- were similar in children, adolescents, and adults. LY900014 demonstrated an accelerated insulin lispro
- absorption with a reduction in the late exposure and an overall shorter PK duration compared to Humalog.
- Following a single subcutaneous bolus infusion with CSII therapy, there was a trend towards an
- accelerated absorption of insulin lispro and the duration of exposure was shorter with LY900014 whilst
- 45 maintaining a similar overall exposure and maximum concentration compared to Humalog in children and
- adolescents with type 1 diabetes (Lilly Internal data).

#### 47 **1.2 Rationale**

52

56

57

64

76

- The rationale for the study is based on the premise that use of an insulin with a more rapid onset of action
- in a CLC system may reduce hyperglycemic excursions, particularly after meals, and may also reduce the
- risk of hypoglycemia due to shorter duration of action. The initial needed determination is that use of
- 51 Lyumjev in the Control-IQ system is safe.

#### 1.3 Potential Risks and Benefits

- Risks and Benefits are detailed below. Loss of confidentiality is a potential risk; however, data are handled
- to minimize this risk. Hypoglycemia, hyperglycemia and ketone formation are always a risk in participants
- with type 1 diabetes and participants will be monitored for these events.

#### 1.3.1 Known Potential Risks

#### **1.3.1.1 Blood Draw**

- A venipuncture and/or fingerstick will be performed to obtain blood for HbA1c measurement.
- Venipuncture can cause common reactions like pain, bruising, or redness at the sampling site.
- 60 Less common reactions include bleeding from the sampling site, formation of a small blood clot or
- 61 swelling of the vein and surrounding tissues, and fainting. A fingerstick frequently causes transient pain
- and there may be a small, localized bruise, which may be followed by a small scar that may persist for
- 63 several weeks. The risk of local infection is less than 1 in 1000 with either venipuncture or fingerstick.

#### 1.3.1.2 CGM and Pump Catheter Risks

- There is a small risk of bleeding where the sensor or infusion set is inserted. There is a small risk for
- developing a local skin infection at the site of CGM sensor placement of pump infusion set placement.
- 67 This may be associated with swelling, redness and pain; and may require antibiotic therapy. Rarely, a
- 68 CGM sensor may break and leave a small portion of the sensor under the skin that may cause redness,
- swelling or pain at the insertion site.
- Nome participants may develop skin irritation or allergic reactions to the adhesives used to secure the
- 71 CGM, or to secure the insulin infusion sets for the continuous subcutaneous insulin infusion. If these
- reactions occur, different adhesives or "under-taping" (such as with IV 3000, Tegaderm, etc.) will be
- tried, sites will be rotated frequently, and a mild topical steroid cream or other medication may be
- required. Skin irritation or allergic reactions at the infusion site could also occur with infusion of
- insulin. As a new insulin is being used in this study, this is a possible risk.

#### 1.3.1.3 Hypoglycemia

- As with any person having type 1 diabetes and using insulin, there is always a risk of having
- hypoglycemia. The frequency of hypoglycemia should be no more and possibly less than it would be
- as part of daily living. Symptoms of hypoglycemia can include sweating, jitteriness, and not feeling well.
- There is the possibility of fainting or seizures (convulsions) and that for a few days the participant may

not be as aware of symptoms of hypoglycemia. A CGM functioning poorly and significantly over-81 reading glucose values could lead to inappropriate insulin delivery. 82

#### 1.3.1.4 Risk of Hyperglycemia

Hyperglycemia and ketonemia could occur if insulin delivery is attenuated or suspended for an extended period or if the pump or infusion set is not working properly. A CGM functioning poorly and significantly under-reading glucose values could lead to inappropriate suspension of insulin delivery.

#### 1.3.1.5 Risk of Device Reuse

The study CGM system is labeled for single use only. The sensor (the component of the system that enters the skin) will be single use only. The receiver, if used, is a hand-held device. The transmitter and receiver may be reused during the study after cleaning the device using a hospital-approved cleaning procedure. The transmitter is attached to the sensor but does not enter the skin. Participants will be informed that FDA or relevant national authorities have approved these devices for single use and that by using them among multiple patients, bloodborne pathogens (i.e. Hepatitis B) may be spread through the use of multiple users.

The study insulin pump is labeled for single-patient use. During the study, this device may be reused 95 96 after cleaning adhering to a hospital-approved cleaning procedure. All infusion set equipment will be 97 single patient use only (infusion set insertion kits, tubing, cartridges etc.) Participants will be informed that FDA or relevant national authorities typically approve the insulin pump device for single use and 98 that by using them among multiple patients, bloodborne pathogens (i.e. Hepatitis B) may be spread 99 through the use of multiple users.

100

83

84

85

86

87

88

89

90

91

92

93 94

104

105

106

107

108

109

110

111

112

113

114

115

116

117

118

101 The study blood glucose meter and blood ketone meter are labeled for single-patient use.

During the study, only one person can use each device as there are rare risks that bloodborne 102

pathogens (i.e. Hepatitis B) may be spread through the use of multiple users. 103

#### 1.3.1.6 Questionnaires

As part of the study, participants (or their parent/legal guardian) will complete questionnaires which include questions about their private attitudes, feelings and behavior related to the investigational equipment as well as managing diabetes. It is possible that some people may find these questionnaires to be mildly upsetting. Similar questionnaires have been used in previous research and these types of reactions have been uncommon.

#### 1.3.1.7 Potential Risks of the CLC System

Even though the study system has been tested prior to this study, there is still a risk that parts of the system may not function properly. The following are possible reasons the system may deliver too much insulin or incorrectly stop insulin delivery:

- CGM sensor reads higher or lower than the actual glucose level which increases risk for hypoglycemia and hyperglycemia with automated insulin delivery system;
- Device malfunctions that could produce a suspension of insulin delivery or over delivery of insulin.

#### 1.3.1.8 Potential Risks of Using Lyumjev

119 Potential adverse reactions with Lyumjev are similar to other insulins: hypoglycemia, hypokalemia, allergic reactions, injection-site reactions, lipodystrophy, localized cutaneous amyloidosis, pruritus, rash, 120

weight gain, and peripheral edema. Infusion site reactions and discomfort will be carefully monitored for in the study.

#### 1.3.1.9 Other Risks

- Data downloaded from the CGM, pump, and the home glucose and ketone meter will be collected for the
- study. The downloaded data from the participant's home pump will include data from prior to the date of
- the screening visit and will include data from the period beyond the last 4 weeks prior to screening. Some
- people may be uncomfortable with the researchers' having such detailed information about their daily
- diabetes habits.

123

129

134

141

#### 1.3.2 Benefits

- Participants may achieve better glucose control than they are currently achieving using the Control IQ
- system. It is expected that this protocol will yield increased knowledge about using the Control-IQ system
- with Lyumjev insulin that will lead to its becoming approved for use.
- The individual participant may not benefit from study participation.

#### 1.3.3 Risk Assessment

- Based on the facts that (1) study participants are already using the Control-IQ system, (2), mitigations
- are in place, and have been tested in prior studies using the investigational device system in the home
- setting, that limit the likelihood of excessive insulin dosing or prolonged withdrawal of insulin, and
- 138 (3) rapid reversal of hypoglycemia and hyperglycemia can be achieved, it is the assessment of the
- investigators that this protocol falls under DHHS 46.405 which is a greater than mimimal risk, but also
- presents prospect of direct benefit to the participants.

#### 1.4 General Considerations

- The study is being conducted in compliance with the policies described in the study policies document,
- with the ethical principles that have their origin in the Declaration of Helsinki, with the protocol
- described herein, and with the standards of Good Clinical Practice (GCP).
- When feasible, data will be directly collected in electronic case report forms, which will be considered
- the source data.
- The protocol is considered a significant risk device study, due to the fact that the intervention is
- experimental. Therefore, an investigational device exemption (IDE) from the U.S. Food and Drug
- Administration (FDA) is required to conduct the study.

# **Chapter 2: Study Enrollment and Lead-in Period**

#### 2.1 Participant Recruitment and Enrollment

- Enrollment will proceed with the goal of having up to 200 participants commencing the treatment period
- so that at least 160 participants complete the trial (approximately 80 participants age 6-<14 years of age,
- and approximately 80 partipants age 14+). At least 20 participants will be age 14-<18 years of age.
- A maximum of 200 individuals may be enrolled into screening (ie, be consented) in the study in order
- to achieve this goal.

151

152

- 158 Study participants will be recruited from ~10-15 clinical centers in the United States without regard to
- gender, race, or ethnicity. There is no restriction on the number of participants to be enrolled by each site
- toward the overall recruitment goal.
- In addition, there will be a study-wide goal to have at least 1/3 of completers with baseline HbA1c  $\geq 7.5\%$ ;
- and at least 10 completers with basal insulin rate >3 units/hour (for at least part of the day).
- 163 Enrollment will be staged, starting with the 14+ cohort. After a cumulative 10,000 hours of use are
- reached in the age 14+ cohort, a Trial Level Safety Review of all adverse events and device issues will be
- performed before opening enrollment to the 6-13 year old cohort. Participants in this review will include
- the Medical Monitor, Sponsor personnel, and a medical representative from Eli Lilly. The decision to
- proceed with enrollment of younger participants will be driven by the totality of the safety data including
- any relevant device or drug
- 169 data.

170

#### 2.1.1 Informed Consent and Authorization Procedures

- Potential eligibility may be assessed as part of a routine-care examination. Before completing any
- procedures or collecting any data that are not part of usual care, electronic informed consent will be
- obtained.
- For potential study participants ≥18 years old, the study protocol will be discussed with the potential
- study participant by study staff. The potential study participant will be given the Informed Consent
- Form to read. Potential study participants will be encouraged to discuss the study with family members
- and their personal physicians(s) before deciding whether to participate in the study. If the potential study
- participant agrees to participate, the Informed Consent Form will be electronically signed through the
- 179 JCHR website.
- For potential participants under 18 years of age, a parent/legal guardian (referred to subsequently as
- "parent") will be provided with the Informed Consent Form to read and will be given the opportunity
- to ask questions. Potential participants meeting the IRB's minimum age of assent will be given a Child
- Assent Form to read and discuss with his/her parents and study personnel. If the parent and child agree
- to participate, the child will provide explicit verbal assent and the Informed Consent Form will be
- electronically signed by the parent through the JCHR website. Both the parent and the Investigator must
- attest that the child provided explicit assent. A failure to object or a lack of response shall not be
- construed to be assent.
- A copy of the consent form (and assent form as applicable) will be provided to the participant or the
- participant and his/her parent and another copy will be added to the participant's study record.
- As part of the informed consent process, each participant/parent will be asked to sign an authorization for
- release of personal information. The investigator, or his or her designee, will review the study-specific
- information that will be collected and to whom that information will be disclosed. After speaking with
- the participant, questions will be answered about the details regarding authorization.

- A participant is considered enrolled when the informed consent form and authorization have been signed
- by all applicable parties.
- Participants who turn 7 during the course of the study will need to read the Child Assent Form and
- provide explicit verbal assent as attested by the parent and Investigator. Participants who turn 18 during
- the course of the study will need to re-consent and provide re-authorization with an adult Informed
- 199 Consent Form.

200

201

205

206

207

208

213

214

215

216

217

218219

220

221

222

223

224

225

226

227

231

#### 2.2 Participant Eligibility Criteria

#### 2.2.1 Inclusion Criteria

- Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study.
- 204 1. Age 6 to <81 years
  - 2. Diagnosis of type 1 diabetes for at least 1 year
  - 3. Currently using Control-IQ technology for at least 3 months, with CGM data recorded indicative of system use (active closed loop) for at least 85% of the possible time in 14 days prior to enrollment
- 4. Total daily insulin dose (TDD) at least 2 U/day
- 210 5. HbA1c < 10.5%
- 6. Residing full-time in the United States, with no anticipated travel outside the United States during the period of study participation.
  - 7. For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact the participant in case of an emergency, and willing to use the Dexcom Follow app (with push notifications turned on) for the duration of the study.
    - 8. If >18 years old, participant has someone who lives within 30 minutes of them who is willing to be contacted if the study team can't reach the participant in case of a suspected medical emergency.
    - 9. Participant has agreed to participate in the study; and has read, understood and signed the informed consent form (ICF) and assent, if applicable; and has agreed to follow all study procedures, including:
      - suspending use of any personal CGM for the duration of the clinical trial once the study CGM is in use
      - switching to or continuing to use Humalog during the lead-in period
  - switching to Lyumjev for the main study period.
  - willing and able to perform the study exercise and meal challenges.
- 10. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, including ability to respond to alerts and alarms, and to provide basic diabetes self-management.
  - 11. Participant and/or parent/legal guardian have the ability to read and understand English

#### 2.2.2 Exclusion Criteria

232

241

2.42 243

244

245

246

247

250

255

256

257

258

259

260

- Individuals meeting any of the following exclusion criteria at baseline will be excluded from study 233 participation. 234
- 1. More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months 235
- 2. More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months 236
- 3. Inpatient psychiatric treatment in the past 6 months 237
- 4. History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to 238 screening or unwillingness to agree to abstain from illicit drugs throughout the study. 239
- 240 5. For Female: Currently pregnant or planning to become pregnant during the time period of study participation
  - A negative pregnancy test will be required for all females of child-bearing potential (menarchal)
  - Counseling on appropriate birth control options will be provided to females with childbearing potential in the event the participant does not have an acceptable plan.
  - 6. Adults lacking the capacity to provide consent and/or follow study procedures in the opinion of the investigator
- 7. Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, 248 GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas). 249
  - 8. Hemophilia or any other bleeding disorder
- 9. Hemoglobinopathy 251
- 10. History of heart, liver, lung or kidney disease determined by investigator to interfere with the 252 study 253
- 11. History of allergic reaction to Humalog or Lyumjev 254
  - 12. Use of glucocorticoids, beta blockers or other medications determined by investigator to interfere with study
    - 13. Abnormal screening electrocardiogram consistent with increased risk during exercise, such as arrhythmia, ischemia, or prolonged QTc interval (>450 ms) (Screening ECG only required for participants age > 50 years, duration of diabetes > 20 years, or history of coronary artery disease)
      - 14. Significant chronic kidney disease (which could impact CGM accuracy in investigator's judgment) or hemodialysis
- 15. History of adrenal insufficiency 262
- 16. History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not 263 appropriately treated 264
- 17. History of gastroparesis 265
- 18. A condition, which in the opinion of the investigator or designee, would put the participant or 2.66 study at risk 267
- 19. Participation in another pharmaceutical or device trial at the time of enrollment or anticipated for 268 during the time period of study participation 269

- 20. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc.,
  Eli Lilly and Co., or TypeZero Technologies, LLC, or having a direct supervisor at place of
  employment who is also directly involved in conducting the clinical trial (as a study investigator,
  coordinator, etc.): or having a first-degree relative who is directly involved in conducting the
- coordinator, etc.); or having a first-degree relative who is directly involved in conducting the
- 274 clinical trial

275

279

290

291

295

296

303

#### 2.3 Screening Procedures

- After informed consent has been signed, a potential participant will be evaluated for study eligibility
- 277 through the elicitation of a medical history, performance of a physical examination by study personnel
- and local laboratory testing if needed to screen for exclusionary medical conditions.

#### 2.3.1 Data Collection and Testing

- A standard physical exam (including vital signs and height and weight measurements) will be performed
- by the study investigator or designee (a physician, fellow, nurse practitioner or a physician assistant).
- The following procedures will be performed/data collected/eligibility criteria checked and documented:
- Inclusion and exclusion criteria assessed
- Demographics (date of birth, sex, race and ethnicity)
- Contact information (retained at the site and not entered into study database)
- Medical history
- Substance use history (drinking, smoking, and drug habits)
- Concomitant medications
- Physical examination to include:
  - Weight, height
  - Vital signs including measurement of blood pressure and pulse
- Blood draw (venipuncture or fingerstick) for local HbA1c measurement
- Urine pregnancy test (test not required for any female that has not reached menarche, is surgically sterile, or is at least 1 year post-menopausal)
  - For those not excluded from testing, counseling on appropriate birth control options will be provided in the event the participant does not have an acceptable plan.
- ECG performed at screening for participants age > 50 years, duration of diabetes > 20 years, or history of coronary artery disease
- Completion of the following patient-reported outcomes (PRO) surveys by the participant (age 14+) or parent: TRIM-D, Trim-DD (Diabetes Device), ITSQ (Insulin Treatment Satisfaction Questionnaire)
- 302 Screening procedures will last approximately 1-2 hours.

#### 2.4 Screen Failures

- Individuals who do not initially meet study eligibility requirements may be rescreened one more time at a
- later date per investigator discretion.

#### 2.5 Lead-in Period

- All participants will complete the Lead-in Period as an outpatient for approximately 16 days. The Lead-in
- Period may begin the same day the screening visit is completed or within 4 weeks after informed consent
- is signed. The lead-in period will last at least 16 days and no more than 21 days.
- At the initiation of the Lead-in Period (CIQ 1.5/ Humalog Training Visit), participants will switch from
- their current Control-IQ system to the study pump (Control-IQ 1.5 technology), study sensor, and study-
- provided Humalog (insulin lispro injection). Training will be provided by qualified study staff on the
- study pump, the study CGM sensor, the study glucose meter, and the study ketone meter. The study
- investigator may adjust insulin delivery profile settings as indicated.
- During the lead-in period, each participant will perform one meal and exercise challenge to determine a
- baseline using Humalog and Control-IQ 1.5. Those day and overnight periods will be analyzed separately.
- Procedures are described in section 5.1. A minimum of 48 hours will occur between all challenges for
- each participant.
- After 16 days (and up to 21 days), the participant will have a visit. System use will be assessed and to
- proceed to the Treatment Period, it is necessary that a participant used the Control-IQ system, with at
- least 85% of system use (active closed loop) reported over the time of the lead-in period (ie, minimum of
- 322 85% of 14 days).
- The lead-in period data collection may be repeated if this threshold is not met.

# **Chapter 3: Treatment Period**

#### 325 3.1 CIQ 1.5/ Lyumjev Training Visit

- At the end of the Lead-in Period, participants will have a clinic visit at which their use of the CIQ 1.5
- 327 system with Humalog will be assessed. Participants who successfully used the system with at least
- 85% of system use (active closed loop) will undergo device training with Lyumjev in the study pump.
- A blood sample (venipuncture or fingerstick) will be obtained to send to the central laboratory for
- 330 HbA1c measurement.

324

333

339

340

341

342

- Participants will receive supplies for blood glucose and ketone testing. QC testing will be performed on
- the meters before they are dispensed.

#### 3.1.1 Training on System Use

- All participants will receive study system training from a qualified trainer. Since all of the participants
- will be experienced Control-IQ users, the amount of training will be customized for each participant.
- For pediatric participants, a parent (or legal guardian) will be required to attend the training procedures.
- At a minimum training will include the following:
- Calibration of the CGM in accordance with manufacturer labeling
  - Use of Lyumjev in the study pump
  - Procedures for treating severe hypoglycemia
  - Procedures for identifying potential infusion set failure and steps to take including the checking of the blood ketone level and changing the infusion set
- The participant will be given a User Guide as a reference as well as Hypoglycemia and Hyperglycemia
- 344 Guidelines.
- Participants will be instructed to download the study device prior to each phone contact or office visit.
- The participant will be instructed to use the system in closed-loop mode except 1) when no calibrated
- CGM sensor is available or 2) if insulin is delivered by any means other than the study pump (e.g.
- injection of subcutaneous insulin via syringe in the event of infusion site failure). If insulin is delivered
- by any means other than the study pump, participant will be instructed to turn off Control-IQ for four
- 350 hours.
- The participant will also be instructed to contact study staff during periods of illness with an elevated
- temperature >101.5 degrees Fahrenheit (38.6 degrees Celsius), periods of significant illness, or during
- periods of use of medications such as epinephrine for the emergency treatment of a severe allergic
- reaction or asthma attack in addition to use of oral or injectable glucocorticoids to determine if closed-
- loop use should be temporarily discontinued.
- Participants will be provided with contact information and will be asked to call the study clinical staff
- for any health-related issues and for technical issues with the system. Participants may use the study
- pump without Control-IQ activated and study CGM during periods of component disconnections or
- 359 technical difficulties.
- Adult participants may use available manufacturer-provided CGM software and features of the study
- CGM related to mobile data access or remote monitoring, but will be instructed not to use any third-party
- components for this purpose. For pediatric participants, the parent/caregiver will use the Dexcom Follow
- app (with push notifications turned on) for the duration of the study.

- The t:connect mobile app from Tandem Diabetes Care will not be available for use during the trial, and
- will not pair to the study pump.

372

386

396

397

398

399

400

401

402 403

404

- Study staff will discuss with the participant that routine contact is required and will make arrangements
- with the participant for the contacts. If the participant cannot be reached, the participant's other contact
- methods will be utilized, including the emergency contact. Participants who are not compliant with the
- arranged contacts on two separate occasions may be discontinued at the discretion of the investigator.
- Following the CIO 1.5/Lyumjey Training Visit, participants will use the study pump and the
- investigational insulin for ~90 days during the Treatment Period.

#### 3.1.2 Training on Management of Hypoglycemia

- The t:slim X2 with Control-IQ system will issue a predictive hypoglycemia alert (Control-IQ Low Alert)
- when the system predicts BG <70 mg/dL within the next 15 minutes (<80 mg/dL when exercise mode is
- activated). Participants will be permitted to change the CGM low glucose threshold alert setting on their
- device or mobile app, but will be instructed to choose a value no less than 70 mg/dL.
- 377 If the participant receives a Control-IQ Low Alert, a message appears on the user interface (UI) that is
- accompanied by vibration followed by vibrations and/or sound if not acknowledged by the user in 5
- minutes. This alert remains on the screen until acknowledged by the participant. The user is prompted
- to test blood glucose and treat with carbohydrate.
- The participant and companion if available will be instructed that if severe hypoglycemia occurs, the
- study pump's insulin delivery should be suspended and glucagon administration if the participant is
- unable to consume carbohydrate.
- Participants will be required to have a home glucagon emergency kit. Participants who currently do not
- have one will be given a prescription for the glucagon emergency kit.

#### 3.1.3 Training on Management of Hyperglycemia

- The t:slim X2 with Control-IO system will issue a predictive hyperglycemia alert (Control-IO High Alert)
- when the system has increased insulin delivery, but detects a CGM value above 200 mg/dL and does not
- predict the value will decrease in the next 30 minutes. During the course of the study, participants will be
- permitted to change the CGM high glucose threshold alert setting on their device or mobile app, but will
- be instructed to choose a value no greater than 300 mg/dL.
- 392 If the participant receives a Control-IQ High Alert, a prompt appears on the user interface to check the
- site for occlusion and test blood glucose.
- 394 If a participant's CGM reading is >300 mg/dL for more than 60 minutes or is ≥400 mg/dL at any point,
- the participant will be instructed to take the following steps:
  - Perform a blood glucose meter check.
    - If the blood glucose is >300 mg/dL, check for blood ketones with the study ketone meter.
    - If the ketone level is ≥ 0.6 mmol/L (or ≥ 2.5 mmol\L at any time), take correction insulin, change insulin (pump) infusion site and contact study staff. Continue to monitor their glucose and blood ketone levels until they return to normoglycemia and ketones are < 0.6 mmol/l.
      - If ketones are <0.6 mmol/l, they will be advised to continue to monitor their glucose until it returns to normoglycemia and to repeat the ketone measurement in 90 minutes if necessary
    - If correction insulin is administered via insulin syringe, turn Control-IQ off for four hours and until glucose level has returned to <180 mg/dL.

#### 3.1.4 Participant Reporting of Infusion Set Insertion Reactions

- Participants will receive a weekly contact (phone, email and/or text message) to assess any issues related to their current infusion site.
- 408 Participants will be instructed to take a photo at time of removal of the first 2 infusion sets and
- subsequently photo at the time of removal only if there is redness on skin when the infusion set is
- removed. Additional photos may be needed if during a virtual visit, video is not available.

#### 3.1.5 Adjustments in Insulin Pump Settings

- Insulin and glucose data from the Lead-in Period will be reviewed and the site investigator may adjust
- 413 insulin delivery profile settings as needed in accordance with their clinical practice.

#### 3.2 Study Visits and Phone Contacts

405

411

414

427

428

429

430

431

432

- Participants will have a phone (or video-conference) follow-up visit at 3 days, 1 week, 2 weeks, and 3
- weeks, a clinic follow-up visit at 6 weeks, a phone follow-up visit at 9 weeks, and a final clinic visit at 13
- weeks, within the windows specified below.

| TARGET<br>DAY/WEEK | VISIT OR<br>PHONE | TARGET WINDOW<br>(AROUND TARGET<br>DAY/WEEK) |
|---|---|---|
| 3 day | P | <u>+</u> 1 day |
| 1 week | P | <u>+</u> 2 days |
| 2 week | P | <u>+</u> 2 days |
| 3 weeks | P | <u>+</u> 7 days |
| 6 weeks | V | <u>+</u> 7 days |
| 9 weeks | P | <u>+</u> 7 days |
| 13 weeks | V | 91-98 days |

- If necessary, visits should be completed out-of-window rather than missed. A visit is not considered
- missed until the next visit/phone window opens.
- The goal will be for all participants to complete all scheduled visits. However, participants who
- (because of unforeseen circumstances or due to changes in contact precautions that may be needed
- during the evolving COVID-19 pandemic) are unable or unwilling to return for all follow-up visits
- will be permitted to return for key visits only as an alternative to withdrawal from the study. When a
- 424 participant is placed into this status, missed visits will not be recorded as protocol deviations (since
- they would not be recorded as protocol deviations if the participant was dropped from the study).
- 426 Additional office visits may occur as needed.

#### 3.2.1 Procedures During Phone Contacts

- Phone contacts can be with or without video. Phone contacts will include the following:
  - Assessment of device issues that have occurred
  - Assessment of adverse events (such as hyperglcyemia, hypoglcyemia, and infusion set reactions)
    using open ended questions, and their underlying cause and relationship to the study device, study
    insulin or other parts of the system (such as the infusion set).

- Completion of a detailed case report form with respect to any infusion site reactions that have occurred.
- For the first three contacts (3 day, 1 week, 2 week), if a video virtual visit can be done, visual inspection
- will be performed of the current and most recent infusion set insertion site. If video is not possible, then
- the participant will be requested to take a photo of the current and most recent infusion set insertion sites.

#### 3.2.2 Procedures at Study Visits

- The following procedures will be performed at each visit, unless otherwise specified:
- Review of study device data
- Assessment of compliance with study device use by review of any available device data
- Assessment of device issues that have occurred
  - Assessment of adverse events, using open ended questions to capture hyperglycemic and hypoglycemic events, and their underlying cause and relationship to the study device, study insulin or other parts of the system (such as the infusion set).
  - A focusesd physical exam to include skin and infusion sites will be performed at each in person visit.
    - Completion of a detailed case report form with respect to any infusion site reactions that have occurred.
- At 13 weeks, the following additional procedures will be performed:
  - Blood draw (venipuncture or fingerstick) for HbA1c measurement at central lab (13 weeks only)
- Completion of the following PRO surveys by the participant (age 14+) or parent: TRIM-D, Trim-DD (Diabetes Device), ITSQ (Insulin Treatment Satisfaction Questionnaire)

#### 3.2.3 Unscheduled Visits

- Participants may have unscheduled visits during the study period if required for additional device training
- or other unanticipated needs per the study investigator discretion.

#### 457 **3.3 Exercise and Meal Challenges**

- 458 Participants will complete 3 meal and 3 exercise challenges during Lyumjev use. Procedures are
- described in section 5.1.

#### 3.4 Early Discontinuation of Study Device

- Participants who discontinue the study device prior to 13 weeks, either by choice or by investigator
- decision, will be asked to come for an end of study visit and then will be dropped from the study.
- 463 If the visit occurs at 6 weeks or after, blood will be drawn for the central-lab HbA1c measurement and
- the PROs will be completed.

465

460

438

443

444

445446

447

448

449

451

# **Chapter 4: Study Devices and Drugs**

#### 467 4.1 Study Devices

466

469

471

474

479

488

489

490

491 492

493

494

495

496

497

498

499

The investigational device (CLC system) includes an insulin pump and a continuous glucose monitor.

#### 4.1.1 Insulin Pump

470 The study system will include the Tandem t:slim X2 with Control-IQ technology.

#### 4.1.2 Continuous Glucose Monitoring

- The study CGM that is part of the CLC system is the Dexcom G6, which includes a transmitter and
- sensors. The CGM sensor will be replaced at least once every 10 days.

#### 4.1.3 Blood Glucose Meter

- The study blood glucose meter is the Contour® NEXT (Ascencia Diabetes Care).
- Blood glucose levels will be measured using the study's blood glucose meter (glucometer) and the
- 477 CGM device will be calibrated if needed using the study glucometer and strips in accordance with the
- 478 manufacturer's labeling.

#### 4.1.4 Ketone Meter

- The study blood ketone meter is the Precision Xtra Blood Glucose and Ketone Monitoring System
- (Abbott Diabetes Care ).
- Blood ketone levels will be measured when needed to evaluate prolonged hyperglycemia. The blood
- glucose meter component of the Precision Xtra device will not be used.

#### **484 4.2 Study Drug**

- The study drug is Lyumjev (insulin lispro-aabc). The drug is a formulation of insulin lispro that includes
- the addition of two excipients, treprostinil and sodium citrate. Treprostinil enhances absorption by local
- vasodilatation without eliciting a systemic effect while citrate further enhances the speed of absorption.

#### Acquisition

Study drug will be shipped by Eli Lilly to the study's central pharmacy for distribution to the clinical sites.

#### • Formulation, Appearance, Packaging, and Labeling

LYUMJEV (insulin lispro-aabc) injection is a sterile, aqueous, clear, and colorless solution for subcutaneous or intravenous administration. Each mL of LYUMJEV U-100 contains 100 units of insulin lispro-aabc and the inactive ingredients: glycerol (12.1 mg), magnesium chloride hexahydrate (1.02 mg), metacresol (3.15 mg), sodium citrate dihydrate (4.41 mg), treprostinil sodium (1.06 mcg), zinc oxide (content adjusted to provide 39 mcg zinc ion), and Water for Injection, USP.

#### • Product Storage and Stability

- Dispense in the original sealed carton with the enclosed Instructions for Use.
- Refrigerate unopened LYUMJEV vials between 36°F to 46°F (2°C to 8°C) until time of use and keep in the original carton to protect from light. Do not freeze or use LYUMJEV if it has been

| 502 | frozen. Do not expose to direct heat. Discard opened or unopened LYUMJEV vials stored at |
|---|---|
| 503 | room temperature below 86°F (30°C) after 28 days. |

Change the LYUMJEV U-100 in the pump reservoir at least every 9 days, or according to the pump user manual, whichever is shorter, or after exposure to temperatures that exceed 98.6°F (37°C).

| 5 | 06 |
|---|----|
| 5 | 07 |

504

505

| | Not i | n-use | In-use | |
|---|---|---|---|---|
| | (Unop | ened) | (Opened) | |
| | Room Temperature Refrigerated | | Room | Refrigerated |
| | (below 86 F [30 C]) | (36 F to 46 F [2 C to | Temperature | (36 F to 46 F [2 C to |
| | | 8 C]) | (below 86 F [30 C]) | 8 C]) |
| 10 mL | 28 days | Until expiration | 28 days | 28 days |
| vial <sup>a,b</sup> | | date | | |

a In-use (opened) vials, whether or not refrigerated, must be used within 28 days.

510511

512

513

514

508

509

#### 4.3 Study Device and Drug Accountability Procedures

Device and drug accountability procedures will be detailed in the clinical center procedures manual.

#### 4.4 Participant Access to Study Device at Study Closure

- Participants will return all investigational study devices and supplies (insulin pump, CGM and related
- supplies, and unused insulin) at their final visit. Participant may keep the study ketone meter and study
- 517 glucometer if these devices are not marked for investigational use only.

b When stored at room temperature, LYUMJEV can only be used for a total of 28 days including both not in-use (unopened) and in-use (opened) storage time.

# **Chapter 5: Testing Procedures and Questionnaires**

#### 5.1 Meal and Exercise Challenges

518

519

525

531

532

533

535

536

537

538

539

540

541

542

543

544

545

546

547

548

549

551

552

553

554

- Participants will complete 1 missed meal bolus and 1 exercise challenge during the Humalog lead-in
- period, then 3 meal and 3 exercise challenges during Lyumjev use.
- A minimum of 48 hours will occur between all challenges for each participant.
- Participants will be instructed to communicate with study staff within one day prior to each challenge to
- review procedures and to have a contact with study staff after the completion of each challenge.

#### **5.1.1 Meal Challenges**

- The same meal should be used for each of the four meal challenges—either lunch or dinner (participant choice).
- For the lead-in phase meal challenge, no bolus will be given for the meal.
- During Lyumjev use, the three meal challenges will consist of:
- No bolus for the meal
  - 50% bolus calculate the bolus dose using the bolus calculator, and deliver half the recommended dose of insulin.
    - Full bolus for the meal based on calculated bolus dose using the bolus calculator.
- For each meal challenge, participants will:
  - 1. Be in a fasting state for two hours prior to consuming the meal and the last manual insulin bolus more than two hours ago.
  - 2. Only begin the meal challenge if the glucose is between 70 mg/dL and 200 mg/dL. Subjects with hyperglycemia > 200mg/dL will reschedule their challenge for another time. If < 70 mg/dL, carbohydrate treatment can be given and then continue.
  - 3. Consume at least 50 grams carbohydrate for the meal. *Each participant will use the same meal for all of their meal challenges in the study. Participants will be encouraged to use the same frozen entrée of their choice for consistency.*
  - 4. Write down the start and end time of eating the meal, as well as the meal content (to include amount of carbohydrate, protein and fat) on the study provided logbook.
  - 5. Not give an additional bolus for up to 3 hours after the meal challenge, unless BG is above 300 mg/dL for more than 1 hour, or symptoms of hyperglycemia develop.
  - 6. Not take additional carbohydrates for up to 3 hours after the meal challenge, unless BG is < 70 mg/dL, or symptoms of hypoglycemia develop.
    - 7. Not exercise for 3 hours after the meal challenge.
- For pediatric participants, caregivers/parents will be instructed to:
  - Be physically present with the participant and monitor CGM glucose during the 3 hours of each meal bolus challenge timeline.
  - Follow the study hypoglycemia and hyperglycemia safety guidelines, as well as the above guidelines for the challenge.

• Be in same residence with the participant for the overnight period after the challenges and to continue to monitor the participant.

#### **5.1.2 Exercise Challenges**

555

556

557

559

563

564

565

566

567

568

569

570

571

572

573

574

575

576

578

579

580

581

582

583

584

585

589

- For each exercise challenge, participants will:
  - 1. Have extra carbohydrate containing snacks and glucagon on hand during and after exercise.
- 2. Per their usual routine and investigator guidance, consider activation of "exercise activity" on the pump up to 45 minutes ahead of actual exercise, to allow for less insulin on board when starting exercise.
  - 3. Consider reducing the last meal bolus prior to exercise as a way to reduce insulin on board and limit hypoglycemia.
    - 4. Perform two hours of exercise, including at least one hour of moderate activity
  - 5. Only begin exercise if CGM glucose is ≥ 120 mg/dL and CGM glucose is not trending downward.
  - 6. Write down the time of last meal and amount and time of last insulin dose, type of exercise performed, as well as the start and stop time of each exercise session in the study logbook (as this may not correlate exactly with exercise activity use on the pump).
  - 7. Stop the exercise challenges at any point for injury or development of new symptoms (development of chest pain/pressure, feeling unwell, development of hypoglycemic symptoms, undue shortness of breath, signs of poor perfusion (leg pain/claudication), or for any other reason.
  - 8. Notify the site within 24 hours after completion of each exercise challenge if they develop new symptoms and review guidance on the need to stop future exercise challenges if any adverse events or new symptoms occurred per clinician judgement based on the severity of symptoms.
- For pediatric participants, caregivers/parents will be instructed to:
  - Be physically present with the participant and monitor CGM glucose during and through 2 hours after the exercise challenge completes.
    - Follow the study hypoglycemia and hyperglycemia safety guidelines, as well as the above guidelines for the challenge.
    - Be in same residence with the participant for the overnight period after the challenges to continue to monitor the participant.

#### 5.2 Laboratory Testing

#### 5.2.1 HbA1c

- HbA1c measurement will be performed locally at the Screening visit.
- An additional blood sample will be obtained (venipuncture or fingerstick) and sent to central lab at the
- 588 CIQ 1.5/Lyumijev Training visit and at the 13-week visit.

#### **5.2.2 Urine Pregnancy**

- Urine pregnancy testing performed locally at clinical site for females of child-bearing potential at the
- Screening visit and anytime pregnancy is suspected.

#### **5.3 Questionnaires**

Questionnaires are completed during Screening and at the time of the 13-week visit. Each questionnaire is described briefly below. Questionnaires will be completed by participants age 14 years and older, and by parent/guardian for younger participants. The procedures for administration are described in the study procedures manual.

Each questionnaire is described briefly below. The procedures for administration are described in the study procedures manual.

| MEASURE | DESCRIPTION |
|---|---|
| Treatment Related Impact Measure of Diabetes (TRIM-D) | 28-item measure with 5 domains assessing treatment burden, daily life, diabetes management, compliance and psychological health. Higher score indicates a better health state |
| Treatment Related Impact Measure of Diabetes Device (TRIM-DD) | 8-item measure with 2 domains assessing Device Bother and Device Function. Higher score indicates a better health state |
| Insulin Treatment Satisfaction Questionnaire (ITSQ) | 22-item measure with a 5-factor structure assessing insulin satisfaction: satisfaction with insulin delivery device, glycemic control, hypoglycemic control, convenience of regimen and lifestyle flexibility. Scores range from 0 to 100 with higher score indicating a better health state |

599

592

597

# Chapter 6: Unanticipated Problem, Adverse Event, and Device Issue Reporting

#### **6.1 Unanticipated Problems**

Site investigators will promptly report to the Coordinating Center on an eCRF all unanticipated problems meeting the criteria below. Sites overseen by the JCHR IRB must report Unanticipated Problems to the IRB within seven calendar days of recognition. For this protocol, an unanticipated problem is an incident, experience, or outcome that meets all of the following criteria:

- Unexpected (in terms of nature, severity, or frequency) given (a) the research procedures that are described in the protocol related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the subject population being studied
- Related or possibly related to participation in the research (possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research)
- Suggests that the research places participants or others at a greater risk of harm than was previously known or recognized (including physical, psychological, economic, or social harm)

The Coordinating Center also will report to the IRB all unanticipated problems not directly involving a specific site such as unanticipated problems that occur at the Coordinating Center or at another participating entity such as a pharmacy or laboratory. These instances must be reported to the JCHR IRB within seven calendar days of recognition. The Director of the Human Research Protection Program (HRPP) will report to the appropriate regulatory authorities to fulfill the obligations of the HRPP if the IRB determines that the event indeed meets the criteria of an Unanticipated Problem requiring additional reporting.

#### **6.2 Adverse Events**

#### 6.2.1 Definitions

- Adverse Event (AE): Any untoward medical occurrence (including laboratory findings) associated with study procedures, the use of a device, biologic in a study participant, including any comparator used, irrespective of the relationship between the adverse event and the device(s) under investigation (referred to as *Adverse Reaction* when caused by a drug).
- 628 <u>Serious Adverse Event (SAE):</u> Any untoward medical occurrence that meets at least one of the following:
  - Results in death.
  - Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event).
  - Requires inpatient hospitalization or prolongation of existing hospitalization.
  - Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions (sight threatening).
  - Is a congenital anomaly or birth defect.
  - Is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the participant or may require medical/surgical intervention to prevent one of the outcomes listed above).

- 639 <u>Suspected Adverse Reaction:</u> any adverse event for which there is a reasonable possibility that the drug
- caused the adverse event. For the purposes of IND safety reporting, 'reasonable possibility' means there
- is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse
- reaction implies a lesser degree of certainty about causality than adverse reaction, which means any
- adverse event caused by a drug (21 CFR 312.32(a)).
- 644 <u>Suspected Unexpected Serious Adverse Reaction (SUSAR):</u> any adverse event considered to be related
- to a drug that is both unexpected and meets criteria for an SAE. *Unexpected* means that the adverse
- reaction is not listed in the investigator brochure or protocol 21 CFR 312.32(a).
- 647 Unanticipated Adverse Device Effect (UADE): Any serious adverse effect on health or safety or any
- life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death
- was not previously identified in nature, severity, or degree of incidence in the investigational plan or
- application (including a supplementary plan or application), or any other unanticipated serious problem
- associated with a device that relates to the rights, safety, or welfare of participants (21 CFR 812.3(s)).
- 652 <u>Adverse Device Effect (ADE):</u> Any untoward medical occurrence in a study participant which the device
- may have caused or to which the device may have contributed (Note that an Adverse Event Form is to be
- completed in addition to a Device Deficiency or Issue Form, unless excluded from reporting as defined in
- 655 section 6.2.2).

673

676

677

678

679

680

- 656 Comparator: Medical device, therapy (e.g. active treatment, normal clinical practice), placebo or no
- treatment, used in the control group in a clinical investigation. (ISO 14155:2020)
- 658 <u>Device Complaints and Malfunctions:</u> A device complication or complaint is something that happens
- to a device or related to device performance, whereas an adverse event happens to a participant. A device
- complaint may occur independently from an AE, or along with an AE. An AE may occur without a
- device complaint or there may be an AE related to a device complaint. A device malfunction is any
- 662 failure of a device to meet its performance specifications or otherwise perform as intended.
- Performance specifications include all claims made in the labeling for the device. The intended
- performance of a device refers to the intended use for which the device is labeled or marketed.
- 665 (21 CFR 803.3). Note: for reporting purposes, sites will not be asked to distinguish between device
- 666 complaints and malfunctions.
- Use Error: User action or lack of user action while using the medical device (3.34) that leads to a
- different result than that intended by the manufacturer or expected by the user. Includes the inability of
- the user to complete a task. Use errors can result from a mismatch between the characteristics of the user,
- user interface, task or use environment. Users might be aware or unaware that a use error has occurred.
- An unexpected physiological response of the patient is not by itself considered a use error. A malfunction
- of a medical device that causes an unexpected result is not considered a use error. (ISO 14155:2020)

#### **6.2.2 Reportable Adverse Events**

- A reportable adverse event includes all events meeting the definition of an adverse event, except for the following:
  - Hypoglycemia and hyperglycemia not meeting the criteria below will not be recorded as adverse
    events unless associated with an Adverse Device Effect or discontinuation of the study device or
    study drug.
  - Skin reactions from sensor or pump infusion set placement are only reportable as everse advents if severe and/or required treatment (see section 6.2.5).

All reportable AEs—whether volunteered by the participant, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means—will be reported on an AE form online. Each AE form is reviewed by the Medical Monitor to assess safety and to verify the coding and the reporting that is required.

#### **6.2.3** Hypoglycemic Events

Hypoglycemia not associated with an Adverse Device Effect or discontinuation of the study device or study drug is only reportable as an adverse event when one of the following criteria is met:

- a hypoglycemic event occurred meeting the following definition of severe hypoglycemia: the event required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or loss of consciousness. These episodes may be associated with sufficient neuroglycopenia to induce seizure or loss of consciousness. If glucose measurements are not available during such an event, neurological recovery attributable to the restoration of glucose to normal is considered sufficient evidence that the event was induced by a low glucose concentration.
- evaluation or treatment was obtained at a health care provider facility for an acute event involving hypoglycemia, or the participant contacted the site and received guidance following the occurrence of an acute event involving hypoglycemia

When a severe hypoglycemia event occurs (as defined above), a Hypoglycemia Form should be completed in addition to the Adverse Event Form. Severe hypoglycemia events should be considered to be serious adverse events with respect to reporting requirements. When a severe hypoglycemia event occurs during use of a study device, it generally will be considered to be unrelated to the device (per section 6.2.6) if the device functioned as intended and there does not appear to be a flaw in how the device is intended to function.

#### **6.2.4** Hyperglycemic/Ketotic Events

Hyperglycemia not associated with an Adverse Device Effect or discontinuation of the study device or study drug is only reportable as an adverse event when one of the following criteria is met:

- the event involved DKA, as defined by the Diabetes Control and Complications Trial (DCCT) and described below
- evaluation or treatment was obtained at a health care provider facility for an acute event involving hyperglycemia or ketosis, or the participant contacted the site and received guidance on how to manage the hyperglycemia/ketosis
- blood ketone level ≥1.0 mmol/L, even if there was no communication with a health care provider at the time of the event
- Hyperglycemic events are classified as DKA if the following are present:
  - Symptoms such as polyuria, polydipsia, nausea, or vomiting;
  - Serum ketones > 1.5 mmol/L or large/moderate urine ketones;
- Either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate (or CO2) <15; and
- Treatment provided in a health care facility
- When a hyperglycemia/ketotic event qualifies as an SAE as defined in section 6.2.1, a Hyperglycemia/
- DKA Form should be completed in addition to the Adverse Event Form. Events meeting DKA criteria
- should be considered to be serious adverse events with respect to reporting requirements. Hyperglycemia
- events not meeting criteria for DKA generally will not be considered as serious adverse events unless one
- of the SAE criteria in section 6.2.1 is met.
- When a hyperglycemia/DKA event occurs during use of a study device, it generally will be considered to
- be unrelated to the device (per section 6.2.6) if the device functioned as intended and there does not
- appear to be a flaw in how the device is intended to function.

#### 6.2.5 Skin Reactions Related to Infusion Set

- When a skin reaction related to the infusion set is considered to be mild or moderate in nature, an infusion
- site reaction case report form will be completed at each scheduled visit and phone contact, or in response
- to the weekly contact from the sites. When a skin reaction related to the infusion set is considered severe
- or treatment was received, an infusion site reaction case report form and an Adverse Event Form also will
- be completed.

730

736

# 6.2.6 Relationship of Adverse Event to Study Investigational Device

- 737 The study investigator will assess the relationship of any adverse event to the study device or study drug.
- The Medical Monitor also will make this assessment, which may or may not agree with that of the study
- investigator. Reporting requirements will be based on the Medical Monitor's assessment.
- To ensure consistency of adverse event causality assessments, investigators should apply the following
- general guidelines when determining whether an adverse event is related to a study device or study drug:
- 742 **Unrelated:** The AE is clearly not related to a study drug/device and a likely alternative etiology exists
- such as an underlying disease, environmental or toxic factors or other therapy.
- 744 **Unlikely Related:** The AE does not follow a reasonable temporal sequence during or after use of study
- drug/device and a more likely alternative etiology exists such as an underlying disease, environmental or
- toxic factors, or other therapy.
- 747 **Possibly Related:** The AE occurred in a reasonable time during or after use of study drug/device; but
- could be related to another factor such as an underlying disease, environmental or toxic factors, or other
- therapy; and there is a possible, though weak, scientific basis for establishing a causal association
- between the AE and the study drug/device.
- 751 **Probably Related:** The AE occurred in a reasonable time during or after use of study drug/device; is
- unlikely to be related to another factor such as an underlying disease, environmental or toxic factors, or
- other therapy; and there is a plausible, though not strong, scientific basis for establishing a causal
- association between the AE and the study drug/device.
- 755 **Definitely Related:** The AE occurred in a reasonable time during or after use of study drug/device;
- cannot be explained by another factor such as an underlying disease, environmental or toxic factors, or
- therapy; and there is a strong scientific basis for establishing a causal association between the AE and the
- study drug/device.

761

- Events determined to be *Possibly Related*, *Probably Related*, or *Definitely Related* will be considered
- 'Related' with respect to any required IRB and FDA reporting.

# **6.2.7** Severity (Intensity) of Adverse Events

- The severity (intensity) of an adverse event will be rated on a three-point scale: (1) mild, (2) moderate,
- or (3) severe. A severity assessment is a clinical determination of the intensity of an event. Thus, a severe

- adverse event is not necessarily serious. For example, itching for several days may be rated as severe, but
- may not be clinically serious.
- MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily
- activities.
- 768 MODERATE: Usually causes a low level of inconvenience, discomfort or concern to the participant
- and may interfere with daily activities, but is usually ameliorated by simple therapeutic measures and
- participant is able to continue in study.
- 771 SEVERE: Interrupts a participant's usual daily activities, causes severe discomfort, may cause
- discontinuation of study device, and generally requires systemic drug therapy or other treatment.

# 6.2.8 Expectedness

- For a serious adverse event that is considered possibly related to study device or drug, the Medical
- Monitor will classify the event as unexpected if the nature, severity, or frequency of the event is not
- consistent with the risk information previously described in the protocol, labeling, or Investigator
- 777 Brochure.

773

778

786

787

788

789

790

791792

793

794795

796

797

798

799 800

801

802

803

# **6.2.9 Coding of Adverse Events**

- Adverse events will be coded using the MedDRA dictionary. To facilitate coding, the site will enter a
- preliminary MedDRA code which the Medical Monitor may accept or change (the Medical Monitor's
- MedDRA coding will be used for all reporting). The Medical Monitor will review the investigator's
- assessment of causality and may agree or disagree. Both the investigator's and Medical Monitor's
- 783 assessments will be recorded. The Medical Monitor will have the final say in determining the causality
- as well as whether an event is classified as a serious adverse event and/or an unanticipated adverse device
- 785 effect.

#### 6.2.10 Outcome of Adverse Events

The outcome of each reportable adverse event will be classified by the investigator as follows:

- RECOVERED/RESOLVED The participant recovered from the AE/SAE without sequelae. Record the AE/SAE stop date.
- RECOVERED/RESOLVED WITH SEQUELAE The event persisted and had stabilized without change in the event anticipated. Record the AE/SAE stop date.
- FATAL A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death.
- NOT RECOVERED/NOT RESOLVED (ONGOING) An ongoing AE/SAE is defined as the event was ongoing with an undetermined outcome.
- An ongoing outcome will require follow-up by the site in order to determine the final outcome of the AE/SAE. The outcome of an ongoing event at the time of death that was not the cause of death, will be updated and recorded as "resolved" with the date of death recorded as the stop date
- UNKNOWN An unknown outcome is defined as an inability to access the participant or the
  participant's records to determine the outcome (for example, a participant that was lost to followup).

- If any reported adverse events are ongoing when a participant completes the study (or withdraws),
- adverse events classified as UADEs or related SAEs or SUSARs will be followed until they are either
- resolved, or have no prospect of improvement or change, even after the participant has completed all
- applicable study visits/contacts. For all other adverse events, data collection will end at the time the
- participant completes the study. Note: participants should continue to receive appropriate medical care
- for an adverse event after their participation in the study ends.

# 6.3 Reportable Device Issues

- All UADEs and ADEs as defined in section 6.2.1 will be reported on both a device issue form and AE
- form, except for skin reactions from CGM sensor placement or pump infusion set placement that do not
- require pharmacologic treatment.

810

817

821

822

825

- Device complaints and device malfunctions will be reported except in the following circumstances.
- These occurrences are expected and will not be reported on a Device Issue Form assuming criteria for
- a UADE or ADE have not been met:
  - CGM sensor lasting fewer days than expected per manufacturer
- CGM tape adherence issues
- Pump infusion set insertion lasting fewer days than expected per manufacturer
- Battery lifespan deficiency due to inadequate charging or extensive wireless communication
  - Intermittent device component disconnections/communication failures not requiring system replacement or workaround/resolution not specified in user guide/manual.
- Device issues clearly addressed in the user guide manual that do not require additional troubleshooting

# 6.4 Timing of Event Reporting

- SAEs possibly related to a study device, study drug, or study participation and UADEs and SUSARs
- must be reported by the investigator to the Coordinating Center within 24 hours of the site becoming
- aware of the event. This can occur via phone or email, or by completion of the online serious adverse
- event form and device issue form if applicable. If the form is not initially completed, it should be
- competed as soon as possible after there is sufficient information to evaluate the event. All other
- reportable ADEs and other reportable AEs should be submitted by completion on the on line form
- within 7 days of the site becoming aware of the event.
- The Coordinating Center will notify all participating investigators of any adverse event that is
- serious, related, and unexpected. Notification will be made within 10 working days after the
- 835 Coordinating Center becomes aware of the event.
- 836 Each principal investigator is responsible for reporting serious study-related adverse events and abiding
- by any other reporting requirements specific to his/her Institutional Review Board or Ethics Committee.
- Where the JCHR IRB is the overseeing IRB, sites must report all serious, related adverse events within
- 839 seven calendar days.
- Upon receipt of a qualifying event, the Sponsor will investigate the event to determine if a UADE has
- occurred, and if indicated, report the results of the investigation to all overseeing IRBs, and the FDA
- within 10 working days of the Sponsor becoming aware of the UADE per 21CFR 812.46(b). A SUSAR
- must be reported within 7 calendar days if life threatening and 15 calendar days if not life threatening per
- 21 CFR 312.32(c)(2). The Sponsor in conjunction with the Medical Monitor must determine if the UADE
- presents an unreasonable risk to participants. If so, the Sponsor must ensure that all investigations, or
- parts of investigations presenting that risk, are terminated as soon as possible but no later than 5 working

- days after the Sponsor makes this determination and no later than 15 working days after first receipt
- notice of the UADE.
- The investigators are also required to report, without unjustified delay, all device deficiencies that could
- have led to a UADE, including device deficiencies, irrespective of whether an adverse event occurred.

# 851 **6.5 Safety Oversight**

- The study Medical Monitor will review all adverse events and adverse device events that are reported
- during the study and assess the relationship to the study device/drug. SAEs typically will be reviewed
- within 24 hours of reporting. Other AEs typically will be reviewed on a weekly basis. Additionally, the
- Medical Monitor will review compiled safety data at periodic intervals.
- The Sponsor will be informed of all reported adverse evens and the Medical Monitor's assessment of
- relationship to the study device/drug; and informed of all reported device issues.

# 6.6 Stopping Criteria

858

859 860

861

862

863

864

867

868

869

870

871

873

## **6.6.1 Participant Discontinuation of Study Device**

- In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or DKA event (or a malfunction that could have led to severe hypoglycemia or DKA), use of the study device will be suspended while the problem is diagnosed. The UADE will be reported to the IRB and FDA. After assessment of the problem and any correction, use of the study device will not be restarted until approval is received from the IRB and FDA.
- In the absence of a device malfunction, use of the study device by a participant will be discontinued if any of the following occur:
  - The investigator believes it is unsafe for the participant to continue on the intervention. This could be due to the development of a new medical condition or worsening of an existing condition; or participant behavior contrary to the indications for use of the device that imposes on the participant's safety
  - The participant requests that the treatment be stopped
- Participant pregnancy
  - Two distinct episodes of DKA as defined in section 6.2.3
- Two distinct severe hypoglycemia events as defined in section 6.2.3
- One episode of DKA as defined in section 6.2.4 and one severe hypoglycemia event as defined in section 6.2.3
- Each DKA, severe hypoglycemia event, or significant infusion site reaction will be reviewed by the
- Medical Monitor and by the Sponsor with respect to determination of cause and whether the occurrence
- of the event can be attributed to use of the study device or study drug.
- An additional requirement for continued study device use following a single DKA or severe
- hypoglycemia event will be that the site investigator believes that the event is unlikely to recur and that
- it is safe for the participant to continue to use the system. Additionally, if the Medical Monitor determines
- that the occurrence of the event indicates that it is not safe for the participant to continue to use the study
- device, use will be discontinued.

# 6.6.2 Criteria for Suspending or Stopping Overall Study

- In addition to the suspension of device use due to a UADE as described in section 6.2.1, study activities 886 could be similarly suspended if the manufacturer of any constituent study device requires stoppage of 887 device use for safety reasons (e.g. product recall). The affected study activities may resume if the 888 underlying problem can be corrected by a protocol or system modification that will not invalidate the 889 results obtained prior to suspension. 890 In addition to the suspension of closed-loop mode use due to a UADE as described above, closed-loop 891 892 system use will be suspended for a root cause analysis if there are 5 or more cases of severe hypoglycemia or five or more cases of hyperglycemia/ketotic events qualifying as SAEs across the entire 893 study in participants who have initiated Control-IQ technology use. 894
- For pediatric participants, the study will be suspended for that cohort for a root cause analysis if there are 3 or more cases of severe hypoglycemia or 3 or more cases of hyperglycemia/ketotic events qualifying as
- SAEs across the pediatric participants who have initiated Control-IQ technology use.

# **Chapter 7: Miscellaneous Considerations**

898

#### 7.1 Drugs Used as Part of the Protocol 899 Humalog (insulin lispro) will be used during the Lead-in Period and Lyumjey (insulin lispro-aabc) will 900 be used during the Treatment Period. 901 7.2 Collection of Medical Conditions and Medications 902 *Pre-Existing Conditions:* Any medical condition that is either present at screening, a chronic disease, 903 or a prior condition that could impact the participant's health during the course of the study (e.g., prior 904 myocardial infarction or stroke) will be recorded. 905 906 Medical Conditions Developing During the Study: Medical conditions that develop or worsen during the study will be recorded as adverse events. 907 *Medications:* All medications for in use at the time of screening or added during the course of the study 908 will be recorded. Nutraceuticals and preventative treatment also will be recorded. Medications only taken 909 as needed either can be recorded when prescribed or only recorded if used during the study. Glucagon for 910 treatment of severe hypoglycemia will only be recorded if used during the study. 911 7.3 Prohibited Medications, Devices, Treatments, and Procedures 912 Treatment with any insulin other than study-provided insulin and treatment with a non-insulin 913 914 glucose-lowering agent, other than metformin, is not permitted, including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas. 915 The investigational study devices (t:slim X2 insulin pump, Dexcom CGM sensor) must be removed 916 before magnetic resonance imaging (MRI), computed tomography (CT) or diathermy treatment. 917 Participants may continue in the trial after temporarily discontinuing use if requiring one of the above. 918 919 7.4 Rescue Medications, Treatments, and Procedures 920 Each participant will be required to have a glucagon preparation for rescue therapy for severe hypoglycemia. 921 7.5 Pregnancy Reporting 922 If pregnancy occurs, the participant will be discontinued from the study. The occurrence of pregnancy 923 will be reported to the Coordinating Center within seven days and to the JCHR IRB as an Unanticipated 924 Problem within seven calendar days. 925 7.6 Participant Compensation 926 Participant compensation will be specified in the informed consent form. 927

Participation in the study is voluntary, and a participant may withdraw at any time. For participants who

withdraw, their data will be used up until the time of withdrawal.

7.7 Participant Withdrawal

928

929

# 7.8 Confidentiality

For security and confidentiality purposes, participants will be assigned an identifier that will be used instead of their name. Protected health information gathered for this study will be shared with the coordinating center, the Jaeb Center for Health Research in Tampa, FL. De-identified participant information may also be provided to research sites involved in the study.

936

# **Chapter 8: Statistical Considerations**

# 938 8.1 Statistical and Analytical Plans

The approach to sample size and statistical analyses are summarized below.

## 8.2 Statistical Hypotheses

- The primary objective of the study is assessment of safety. Therefore, there is no formal statistical
- hypothesis testing for efficacy. Safety endpoints will be compared with historical published data.

## **8.3 Sample Size**

937

940

946

948

954

955

957

958

961

962

- The sample size of 160 completers of the trial was selected to have reasonable precision for assessing
- safety endpoints and is not based on statistical principles.

#### 8.4 Outcome Measures

## 947 Key Safety Endpoints

- Severe hypoglycemia as defined in section 6.2.3
- Diabetic ketoacidosis as defined in section 6.2.4
- Unanticipated adverse device effects
- Other serious adverse events
- Adverse drug reactions

#### 953 Secondary Safety Endpoints

- All reportable adverse events
  - CGM hypoglycemia outcomes
- Overall % time <54 mg/dL
  - Postprandial % time <54 mg/dL (30 min, <1, <2, <4, >1 to <2 and >2 to <4hr)
  - Overall and postprandial % time <70 mg/dL
- Rate of hypoglycemia events defined as 15 or more consecutive minutes <54 mg/dL

#### 960 Exploratory Endpoints

- Postprandial incremental area under the glucose curve (4 hr)
- Peak postprandial glucose
- Times in ranges-overall and postprandial (70-180 mg/dL, >180 mg/dL, >250 mg/dL, 70-140 mg/dL)
- Mean glucose
- Rate of hyperglycemia events, defined as 90 or more minutes >300 mg/dL within 120 minutes
- Overall variability (CV and SD)
- HbA1c change from baseline
- CGM metrics for hypoglycemia, hyperglycemia, and variability during daytime and nighttime

### Patient-Reported Outcomes

971 • TRIM-D

970

974

982

983

995

1006

- 972 Trim-DD
- 973 ITSO

# 8.5 Analysis Datasets

- For the main analyses, adult and pediatric participants will be pooled. Secondarily separate analyses will
- be conducted for adults (>18 years) and pediatric (<18 years) participants. Further exploratory analyses
- will be conducted within pediatric subgroups.
- All participants who initiate the Treatment Period and use the study device with the study drug will be
- 979 included in the safety analyses.
- For inclusion in the analysis of CGM metrics, participants must have at least 24 hours of CGM data
- during the Treatment Period.

#### 8.6 Statistical Methods

# 8.6.1 Analysis of the Safety Event Endpoints

- Safety events (ie, not including CGM defined events) will be tabulated for each type of event as the
- number of events per participant, the number of participants with > 1 event, and the rate of events per
- 986 100 person-years.
- 987 Since study eligibility excluded participants with 2 or more severe hypoglycemia or DKA events in the
- prior 6 months, an unbiased comparison of the event rate during the Treatment Period with the pre-study
- event rate is not possible. Therefore, the severe hypoglycemia and DKA event rates will be compared
- 990 with the T1D Exchange data. which reported the frequency of 1 or more severe hypoglycemia and DKA
- events in the prior 3 months according to age group; this will allow for age-matching with this trial. The
- proportion of participants with events during the Treatment Period will be compared with the T1D
- 993 Exchange frequency using Barnard's exact test. Study endpoint will be met if severe hypoglycemia and
- DKA event rates are not significantly higher during follow-up compared with T1D Exchange frequency.

# 8.6.2 Analysis of CGM Endpoints

- 996 CGM metrics will be computed for (1) 4 weeks pre-study (personal CGM), (2) Lead-in Period, and
- 997 (3) Treatment Period. CGM metrics will be computed over 24 hours, during daytime (6am-11:59pm),
- during nighttime (12mn-5:59am), and during scheduled exercise and meal challenges.
- The main statistical comparison will be made between the Treatment Period and the Lead-in Period. The
- lead-in period time for analysis will exclude the day and night of the baseline exercise and meal
- 1001 challenges. Additionally the Treatment Period will be compared with the pre-study CGM data.
- Linear mixed models will be used to test the change from pre-Treatment Period to Treatment Period.
- 1003 Missing data will be handled by the method of direct likelihood, which assumes outcomes are missing at
- random and estimates follow-up values via maximimum likelihood. Sensitivity analyses will be
- performed to assess the robustness of the results under different missing data assumptions.

#### 8.6.3 Analysis of HbA1c and PRO Measures

- Linear mixed models will be used to test the change in HbA1c and PRO scores from baseline to
- 1008 13 weeks. Missing data will be handled by the method of direct likelihood, which assumes outcomes are
- missing at random and estimates follow-up values via maximimum likelihood.

### 1010 **8.7 Intervention Adherence**

- The following tabulations will be performed:
- Sensor use–percent time of use
- Closed loop system use–percent time of use
- % time in different operational modes

### **8.8 Protocol Adherence and Retention**

- The following tabulations and analyses will be performed to assess protocol adherence for the study:
- Number of protocol deviations
- Flow chart accounting for all enrolled participants
- Number of and reasons for unscheduled visits and phone calls
- Number of participants who were enrolled but did not enter the Treatment Period and reasons
- Number of participants who stopped treatment and reasons

# 8.9 Baseline Descriptive Statistics

- Baseline demographic and clinical characteristics of the cohort of participants who initiate the Treatment
- Period will be summarized in a table using summary statistics appropriate to the distribution of each
- variable. Descriptive statistics will be displayed by treatment group for the following:
- 1026 Age

1022

1036

- 1027 Sex
- Race/Ethnicity
- Socio-economic factors (income, education, and/or insurance status)
- Diabetes duration
- 1031 HbA1c
- 1032 BMI
- Total daily insulin
- Prior severe hypoglycemia and DKA events
- Baseline CGM metrics

# 8.10 Additional Tabulations and Analyses

- The following data will be tabulated at baseline and at or over 13 weeks
- Insulin metrics (units/kg): total daily insulin, total daily basal insulin, total daily bolus insulin (plus total daily manual bolus, total daily automated bolus)
- 1040 Weight
- Number and type of infusion set reactions

### **8.11 Device Issues**

- The following tabulations will be performed with respect to device issues:
- Reported device issues according to type of issue

# **8.12 Planned Interim Analyses**

No formal interim analyses are planned.

# **8.13 Subgroup Analyses**

- 1048 Results will be tabulated according to age group, HbA1c, and total daily insulin. Additional subgroups
- will be defined in the Statistical Analysis Plan.

# 1050 8.14 Multiple Comparison/Multiplicity

- Safety event endpoints will not be corrected for multiple comparisons. For CGM, HbA1c, and PRO
- endpoint analyses, the false discovery rate will be controlled using the adaptive Two Stage Group
- Benjamini-Hochberg (TST GBH) method.<sup>6,7</sup>

# **8.15 Analysis of Meal and Exercise Challenges**

- The meal and exercise challenges will be analyzed with the same CGM metrics and safety outcomes
- above to be tabuled during, 2 hours after and overnight for each challenge, and will be detailed in the
- statistical analysis plan. Separate analysis will be conducted for each type of challenge.

# **Chapter 9: Data Collection and Monitoring**

# 9.1 Case Report Forms and Other Data Collection

- The main study data are collected on electronic case report forms (eCRFs). When data are directly
- collected in electronic case report forms, this will be considered the source data. For any data points
- for which the eCRF is not considered source (e.g. lab results that are transcribed from a printed report
- into the eCRF), the original source documentation will be maintained in the participant's study chart
- or medical record. This source must be readily verifiable against the values entered into eCRF.
- Even where all study data are directly entered into the eCRFs at office visits, evidence of interaction
- with a live subject must be recorded (e.g., office note, visit record, etc.).
- Electronic device data files are obtained from the study software and individual hardware components.
- These electronic device files are considered the primary source documentation.
- HbA1c measurements will be made by the central laboratory and the data will be transmitted to the
- 1070 Coordinating Center.

1058

1059

1071

1082

# 9.2 Study Records Retention

- Each participating site will maintain appropriate medical and research records for this trial, in
- compliance with ICH E6 and regulatory and institutional requirements for the protection of
- 1074 confidentiality of participants.
- Study documents should be retained for a minimum of 2 years after the last approval of a marketing
- application in an ICH region and until there are no pending or contemplated marketing applications in an
- 1077 ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development
- of the investigational product. These documents should be retained for a longer period, however,
- if required by local regulations. No records will be destroyed without the written consent of the sponsor,
- if applicable. It is the responsibility of the sponsor to inform the investigator when these documents no
- longer need to be retained.

## 9.3 Quality Assurance and Monitoring

- Designated personnel from the Coordinating Center will be responsible for maintaining quality
- assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is
- conducted and data are generated, documented and reported in compliance with the protocol, Good
- 1086 Clinical Practice (GCP) and the applicable regulatory requirements, as well as to ensure that the rights
- and wellbeing of trial participants are protected and that the reported trial data are accurate, complete,
- and verifiable. Adverse events will be prioritized for monitoring.
- A risk-based monitoring (RBM) plan will be developed and revised as needed during the course of
- the study, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations —
- 1091 A Risk Based Approach to Monitoring" (August 2013). Study conduct and monitoring will conform
- with 21 Code of Federal Regulations (CFR) 812. This plan describes in detail who will conduct the
- monitoring, at what frequency monitoring will be done, at what level of detil monitoring will be
- performed, and the distribution of monitoring reports.
- The data of most importance for monitoring at the site are participant eligibility and adverse events.
- Therefore, the RBM plan will focus on these areas. As much as possible, remote monitoring will be
- performed in real-time with on-site monitoring performed to evaluate the verity and completeness of
- the key site data. Elements of the RBM may include:

Qualification assessment, training, and certification for sites and site personnel 1099 Oversight of Institutional Review Board (IRB) coverage and informed consent procedures 1100 Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review 1101 of entered data and edits, statistical monitoring, study closeout 1102 On-site monitoring (site visits): source data verification, site visit report 1103 1104 Agent/Device accountability Communications with site staff 1105 Patient retention and visit completion 1106 1107 Quality control reports Management of noncompliance 1108 Documenting monitoring activities 1109 Adverse event reporting and monitoring 1110 Coordinating Center representatives or their designees may visit the study facilities at any time in order 1111 to maintain current and personal knowledge of the study through review of the records, comparison 1112 with source documents, observation and discussion of the conduct and progress of the study. 1113 The investigational site will provide direct access to all trial related sites, source data/documents, and 1114 reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory 1115 authorities. 1116

#### 9.4 Protocol Deviations

- A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure requirements. The noncompliance may be either on the part of the participant, the investigator, or the study site staff. A significant (or major) deviation is any deviation that departs from the established materials in such a way that it poses an increase in the risk to subjects, adversely affects the welfare, rights, or safety of the research subjects, or negatively influences the scientific study integrity. As a result of a significant deviation, a corrective and preventive action plan shall be developed by the site and implemented promptly.
- The site PI/study staff is responsible for knowing and adhering to their IRB requirements. Further details about the handling of protocol deviations will be included in the monitoring plan.

1127

# **Chapter 10: Ethics/Protection of Human Participants**

### 10.1 Ethical Standard

- The investigator will ensure that this study is conducted in full conformity with Regulations for the
- Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 CFR
- 1132 Part 56, and/or the ICH E6.

1128

1129

1133

1140

1141

#### 10.2 Institutional Review Boards

- The protocol, informed consent form(s), recruitment materials, and all participant materials will be
- submitted to the IRB for review and approval. Approval of both the protocol and the consent form must
- be obtained before any participant is enrolled. Any amendment to the protocol will require review and
- approval by the IRB before the changes are implemented to the study. All changes to the consent form
- will be IRB approved; a determination will be made regarding whether previously consented participants
- need to be re-consented.

#### 10.3 Informed Consent Process

### 10.3.1 Consent Procedures and Documentation

- Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study
- and continues throughout the individual's study participation. Extensive discussion of risks and possible
- benefits of participation will be provided to the participants and their families. Consent forms will be
- IRB-approved and the participant will be asked to read and review the document. The investigator will
- explain the research study to the participant and answer any questions that may arise. All participants
- will receive a verbal explanation in terms suited to their comprehension of the purposes, procedures,
- and potential risks of the study and of their rights as research participants. Participants will have the
- opportunity to carefully review the written consent form and ask questions prior to signing.
- The participants should have the opportunity to discuss the study with their surrogates or think about
- it prior to agreeing to participate. The participant will sign the informed consent document prior to any
- procedures being done specifically for the study. The participants may withdraw consent at any time
- throughout the course of the trial. A copy of the informed consent document will be given to the
- participants for their records. The rights and welfare of the participants will be protected by emphasizing
- to them that the quality of their medical care will not be adversely affected if they decline to participate
- in this study.

1157

## 10.3.2 Participant and Data Confidentiality

- Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the
- sponsor(s) and their agents. This confidentiality is extended to cover testing of biological samples and
- genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol,
- documentation, data, and all other information generated will be held in strict confidence. No information
- concerning the study or the data will be released to any unauthorized third party without prior written
- approval of the sponsor.
- The study monitor, other authorized representatives of the sponsor, representatives of the IRB, regulatory
- agencies or company supplying study product may inspect all documents and records required to be
- maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital)
- and pharmacy records for the participants in this study. The clinical study site will permit access to such
- 1168 records.

| 1169 | The study participant's contact information will be securely stored at each clinical site for internal use |
|---|---|
| 1170 | during the study. At the end of the study, all records will continue to be kept in a secure location for as |
| 1171 | long a period as dictated by the reviewing IRB, institutional policies, or sponsor requirements. |
| 1172 | Study participant research data, which is for purposes of statistical analysis and scientific reporting, will |
| 1173 | be transmitted to and stored at the Coordinating Center. This will not include the participant's contact or |
| 1174 | identifying information, unless otherwise specified in the informed consent form. Rather, individual |
| 1175 | participants and their research data will be identified by a unique study identification number. The study |
| 1176 | data entry and study management systems used by clinical sites and by the Coordinating Center research |
| 1177 | staff will be secured and password protected. At the end of the study, all study databases will be de- |
| 1178 | identified and archived at the Coordinating Center. |
| 1179 | 10.3.3 Future Use of Stored Specimens and Data |
| 1180 | Data collected for this study will be analyzed and stored at the Coordinating Center. After the study is |

- Data collected for this study will be analyzed and stored at the Coordinating Center. After the study is completed, a dataset will be provided to the study Sponsor.
- No biologic specimens will be stored.

# **Chapter 11: References**

1185

- Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM,
   Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ 3rd, Anderson SM, Church MM,
   Dadlani V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, Beck RW; iDCL
   Trial Research Group. Six-month randomized, multicenter trial of closed-loop control in
   type 1 diabetes. N Engl J Med. 2019; 381:1707-1717.
- Breton MD, Kanapka LG, Beck RW, Ekhlaspour L, Forlenza GP, Cengiz E, Schoelwer M,
   Ruedy KJ, Jost E, Carria L, Emory E, Hsu LJ, Oliveri M, Kollman CC, Dokken BB,
   Weinzimer SA, DeBoer MD, Buckingham BA, Cherñavvsky D, Wadwa RP; iDCL Trial
   Research Group. A randomized trial of closed-loop control in children with type 1 diabetes.
   N Engl J Med. 2020 Aug 27;383(9):836-845.
- 3. Breton M, Kovatchev B. One year real-world use of the Control-IQ advanced hybrid closed loop technology. Diabetes Technol Ther 2021 Published Online:21 Apr 2021 <a href="https://doi.org/10.1089/dia.2021.0097">https://doi.org/10.1089/dia.2021.0097</a>
- Leohr J, Dellva MA, Carter K, LaBell E, Linnebjerg H. Ultra Rapid Lispro (URLi)
   Accelerates Insulin Lispro Absorption and Insulin Action vs Humalog® Consistently Across
   Study Populations: A Pooled Analysis of Pharmacokinetic and Glucodynamic Data. Clin
   Pharmacokinet. 2021 May 27; doi: 10.1007/s40262-021-01030-0. Epub ahead of print.
- 5. Foster et al. State of type 1 diabetes management and outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther 2019; 21: 66-72.
- 6. Benjamini YB, Yekutieli D: The control of the false discovery rate in multiple testing under dependency, 2001; *Ann Stat*, 29(4):1165-1188.
- 7. Hu JX, Zhao H, Zhou HH: False discovery rate control with groups. *J Am Stat Assoc*, 2010; 105(491):1215-1227.